CLINICAL TRIAL: NCT00475163
Title: Mentors in Motion: A Physical Activity Intervention for Obese Adolescents
Acronym: MIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Laurent Legault,MD, MUHC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PED-04-018
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Last update posted 2009-03-04 (Estimated); Status verified 2009-03

CONDITIONS: Obesity
Keywords: Obesity; Mentoring; Fitness; Self-esteem
MeSH Terms: conditions — Obesity | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Behavior modification

SUMMARY:
Assesing the impact of mentoring on the lifestyle choices of adolescents who are overweight

DETAILED DESCRIPTION:
Randomized controlled trial of the impact of weekly contacts with mentors to improve physical activity pattern, self esteem, and weight loss in obese teenagers over a 6 month period.

ELIGIBILITY:
Inclusion Criteria:

* 13-17 yo Able to participate in physical activity

Exclusion Criteria:

* On medications that could affect weight

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2004-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Weight gain
Fitness
self esteem

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Legault, MD, Principal Investigator — Montreal Children's Hospital of the MUHC
Locations (1):
- Montreal Children's Hospital, Montreal, Quebec, Canada